CLINICAL TRIAL: NCT06902311
Title: Ultra Hypo-fractionated Adjuvant Whole Breast Radiation Therapy With Simultaneous Integrated Boost for Early-Stage Breast Cancer (H-ASSIST)
Acronym: H-ASSIST
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC2404
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer; Early-stage Breast Cancer; Ductal Carcinoma in Situ; DCIS
Keywords: whole breast irradiation; WBI; simultaneous integrated tumor bed boost (SIB); SIB; Concurrent boost; adverse effects; toxicity; Radiation-specific toxicity; patient reported outcome; PRO-CTCAE
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- WBI-SIB (Experimental): Five-fraction whole breast irradiation (WBI) with simultaneous integrated tumor bed boost (SIB).
  Interventions: Radiation: Breast Radiotherapy

INTERVENTIONS:
Radiation: Breast Radiotherapy — The tumor bed boost when given at the same time (called a simultaneous integrated boost, SIB) with whole breast irradiation (WBI).

SUMMARY:
This study evaluates the rates of radiation-specific toxicity, quality of life, and oncologic outcomes for early-stage breast cancer and ductal carcinoma in situ treated with 5-fraction whole breast irradiation (WBI) with a simultaneous integrated tumor bed boost (SIB). SIB refers to the technique tumor bed boost given at the same time as standard radiation therapy.

The FAST-Forward trial previously showed that a 1-week course of radiotherapy had similar effects to the traditional 3-week course for early-stage breast cancer after surgery. Given these favorable results, a 5-fraction WBI regimen is appealing for many patients who wish to minimize the number of treatment visits while still reducing their risk of recurrence. Generally, tumor bed boosts further decrease the risk of recurrence, but in the setting of 5-fraction WBI, a more traditional sequential boost technique is utilized.

DETAILED DESCRIPTION:
Multiple recent studies demonstrate the noninferiority of a simultaneous integrated boost (SIB) approach. This study will include women aged 50 years and older who are recommended to receive whole breast irradiation with a standard dose boost and without regional nodal irradiation.

Radiation therapy will consist of 5 fractions delivered every other day (excluding weekends), with a total dose of 26 Gy to the whole breast and a simultaneous integrated boost to a total dose of 30 Gy to the lumpectomy cavity.

The primary outcome of this study is to investigate the rate of moderate to marked adverse effects in the breast and chest wall of patients receiving five-fraction whole-breast radiation therapy with a concurrent boost. Radiation-specific toxicity outcomes will be assessed by clinicians and patients at 12 months, along with evaluations of quality of life and oncologic control at 24 months following treatment.

It is hypothesized that 5-fraction whole breast irradiation with a simultaneous integrated boost will result in clinically acceptable rates of moderate to marked toxicity relative to historical controls, while providing good quality of life and high rates of disease control.

ELIGIBILITY:
In order to participate in this study a subject must meet all of the eligibility criteria outlined below.

Inclusion Criteria:

* Willing and able to provide written informed consent obtained to participate in the study and HIPAA authorization for release of personal health information.
* Women ≥ 50 years of age with confirmed de novo invasive carcinoma of breast or ductal carcinoma in situ.
* Subjects with completed breast-conserving surgery (BCS) with or without sentinel lymph node biopsy (SLNB) or axillary lymph node dissection (ALND).
* Subjects planned to receive either SOC whole breast 3D conformal radiation therapy (3D CRT) or SOC whole breast intensity modulated radiation therapy (IMRT) with standard dose tumor bed boost.
* Subjects with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial, per the discretion of the treating radiation oncologist.
* Enrollment in another clinical trial is allowed if there is no interference with interventions on this trial per discretion of the Principal Investigator.

Exclusion Criteria:

* Receipt of concurrent breast reduction involving tissue rearrangement in the lumpectomy cavity (so that boost cannot be accurately targeted).
* Synchronous bilateral breast cancer requiring bilateral radiation therapy.
* Clinical or imaging evidence of distant metastases.
* Prior ipsilateral breast or thoracic radiation.
* Autoimmune conditions
* Collagen Vascular Disease (such as systemic lupus erythematosus, scleroderma, dermatomyositis, among others)
* Patients with pT4 tumors.
* Patients recommended to receive regional nodal irradiation with associated radiation risks

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Rate of any moderate-marked adverse effects | 1 year
  The rate of moderate to marked adverse effects in the breast or chest wall at 1 year will be measured using a questionnaire called the Clinician Assessment of Radiation-Specific Toxicity by clinican. This will be compared against historical controls. The questionnaire includes 10 items: 4 Likert-type questions and 6 yes/no questions. Items are rated from 0 to 4, with higher scores indicating more adverse effects. A "yes" response indicates the occurrence of an adverse event.

SECONDARY OUTCOMES:
In-breast tumor recurrence | 2 years
  In-breast tumor recurrence at 2 years is defined according to the standard definition as the time from enrollment to any of the following events: invasive ipsilateral recurrence and/or ipsilateral DCIS recurrence.
  Recurrence will be measured via medical record abstraction and clinical evaluation.
Quality of life at measured by European Organization for Research and Treatment of Cancer ( EORTC QLQ-C30) | 12 months
  Quality of life at 12 months will be measured as defined by European Organization for Research and Treatment of Cancer ( EORTC QLQ-C30). The EORTC QLQ-C30 is a cancer-specific instrument with 30 questions that incorporates 9 multi-item scales: 5 functional scales (physical, role, cognitive, emotional, and social); 9 symptom scales (fatigue, pain, nausea and vomiting, dyspnea, insomnia, appetite loss, constipation, diarrhea and financial difficulties); and a global health and quality-of-life scale. Most questions used 4 point scale (1 'Not at all' to 4 'Very much'); 2 questions used 7-point scale (1 'very poor' to 7 'Excellent'). The scores of these scales were averaged from the scores of the component items, transformed and analyzed on a 0 - 100 scale. A higher score=better level of functioning or greater degree of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Dana Casey, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical trials at UNC Lineberger — http://unclineberger.org/patientcare/clinical-trials/clinical-trials